CLINICAL TRIAL: NCT06298604
Title: Comparison Between a Novel Motorized EUS Guided Fine Needle Biopsy (FNB) With Standard Needle for Pancreatic and Liver Biopsies
Brief Title: Motorized Fine Needle Biopsy vs Standard Needles
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Ecuatoriano de Enfermedades Digestivas (Other)
Responsible Party: Principal Investigator, Carlos Robles-Medranda, Head of the Endoscopy Division, Instituto Ecuatoriano de Enfermedades Digestivas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: IECED-12112023
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Pancreas Disease; Liver Diseases
Keywords: Fine-needle biopsy; Endosonography; liver; pancreas; pathology
MeSH Terms: conditions — Pancreatic Diseases; Liver Diseases

STUDY DESIGN:
Intervention Model Description: Prospective, diagnostic,, cross-sectional study
Who Masked: Care Provider
Masking Description: Single masking, the pathologist will be blinded to the needle used for sample collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard EUS-guided FNB (Active Comparator): Patients scheduled for EUS-guided liver or pancreas biopsy will undergo the procedure using a standard 19-gauge needle
  Interventions: Device: EUS-guided standard fine needle biopsy
- Motorized EUS-guided FNB (Experimental): Patients scheduled for EUS-guided liver or pancreas biopsy will undergo the procedure using a motorized 20-gauge needle.
  Interventions: Device: EUS-guided motorized fine needle biopsy

INTERVENTIONS:
Device: EUS-guided standard fine needle biopsy — Using the echoendoscope, a pancreatic lesion or liver parenchyma will be identified, and a 19-gauge standard fine needle biopsy device (Boston Scientific, USA) is inserted on it to obtain the sample or specimen.
  Arms: Standard EUS-guided FNB
Device: EUS-guided motorized fine needle biopsy — Using the echoendoscope, a pancreatic lesion or liver parenchyma will be identified, and a 20-gauge motorized fine needle biopsy device (Limaca, Israel) is inserted on it to obtain the sample or specimen.
  Arms: Motorized EUS-guided FNB

SUMMARY:
Recent improvements in punctures techniques and needles now allow for the collection of high-quality specimens comparable to core needle biopsy. A newly developed motorized fine needle biopsy (mFNB), the Precision-GI (Limaca, Israel) promises intact tissue acquisition without sample damage, relying on controlled axial tissue cutting and high-speed rotational coring for optimized tissue acquisition.

Given the advancement mentioned, the investigators aim to compare the performance of the mFNB with the standard needle during the acquisition of endoscopic ultrasound (EUS)-guided pancreatic and liver specimens through a prospective, interventional, single-center trial. The study will consist of two groups of patients: one assigned to the standard fine needle biopsy (FNB) and the other to the mFNB. The primary study outcomes will include sample quality (core integrity), and diagnostic accuracy.

DETAILED DESCRIPTION:
The development of Endoscopic ultrasound-guided tissue acquisition (EUS-TA) has been remarkable. Initially focused on obtaining samples from the pancreas, it has expanded significantly to include various organs adjacent to the gastrointestinal system (i.e., liver, lymph nodes, adrenal glands).

One of the key advancements in EUS-TA involves the shift from cytological analysis, with fine-needle aspiration (FNA), to histological and even genetic evaluations, with fine-needle biopsies (FNB). FNB addresses some limitations associated with FNA, such as low tumor cellularity and the inability to retain cellular architecture.

Recent improvements in puncture techniques and needles, allow for the collection of high-quality specimens, comparable to core needle biopsy, to achieve standards for specimen adequacy (i.e., intact liver cores of at least 15-20 mm with a complete portal triad count of 11). Some current available needle designs include the crown type, flanged type, 20 Gauge FNB needles with forward-faced core traps, and the fork-tip needles, demonstrating high diagnostic accuracy and a low rate of adverse events.

The Precision-GI is a new motorized fine needle (mFNB) developed by LIMACA Medical in Israel for EUS-guided FNB. It operates using a battery-powered motor that enables controlled axial tissue cutting and high-speed rotational coring for optimized tissue acquisition. Moreover, a sharp stylet facilitates crossing through the gastrointestinal wall, allowing for the reach of target lesions. The rotational electromechanical cutting movement into the lesion promises intact motorized tissue acquisition without sample damage.

In the present study, the investigators aim to compare the performance of the mFNB with the standard needle during the acquisition of EUS-guided pancreatic and liver specimens. The study will consist of two groups of patients: one assigned to the standard fine needle biopsy (FNB) and the other to the mFNB. The primary study outcomes will include sample quality (core integrity), and diagnostic accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 99 years
* Patients referred to our center who require EUS-guided liver or pancreas biopsy.
* Male or female patients.
* Patients able to give consent

Exclusion Criteria:

* Pregnancy or nursing
* Patients with coagulation disorders (platelets <50.000/mm3, international normalised ratio (INR) >2)
* Any underlying medical condition that contraindicates EUS-guided fine needle biopsy such as anatomical alterations, significant gastric outlet obstruction, collateral intervening vessels.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12-09 (Actual); Primary Completion 2024-10-09 (Estimated); Study Completion 2024-12-09 (Estimated)

PRIMARY OUTCOMES:
Endoscopic ultrasound fine needle biopsy sample quality | Up to two hours after the procedures
  Based on tissue "core"; Tissue core is defined as a architecturally intact piece of at least 550 micron in the greatest axis. The tissue core will be evaluated in both groups by the pathologist immediately after its acquisition.
Diagnostic accuracy according to histological analysis | Up to one week
  Proportion of subjects with a definitive diagnosis based on the number of passes and throws for tissue acquisition.

SECONDARY OUTCOMES:
Tissue blood contamination | Up to one hour
  Evaluation of tissue blood contamination will be based on a sample quality score:
  1. Only blood
  2. High (>50% of the surface of the slide)
  3. Moderate (25%-50% of the surface of the slide)
  4. Low (<25% of the surface of the slide)

OTHER OUTCOMES:
Time efficiency during tissue acquisition | Up to two hours
  The tissue from identifying the lesion to obtaining the sample. It will be calculated in minutes
Rate of liver specimen adequacy | Up to 1 week
  Intact liver cores of at least 15-20 mm with a complete portal triad count of 11
Rate of adverse events associated with the procedure | Up to 6 months
  Adverse event associated with the procedure, including transprocedural, early, and late post-procedural occurrence
Quality of cytologic sample | Up to 2 hours
  The quality of the cytologic sample will be scored according to the pathologist criteria as:
  0= insufficient material for cytologic interpretation
  1. sufficient material for limited cytologic interpretation
  2. sufficient material for adequate cytologic interpretation

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Ecuatoriano de Enfermedades Digestivas (IECED), Guayaquil, Ecuador

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mendoza Ladd A, Casner N, Cherukuri SV, Garcia C, Padilla O, Dwivedi A, Hakim N. Fine Needle Biopsies of Solid Pancreatic Lesions: Tissue Acquisition Technique and Needle Design Do Not Impact Specimen Adequacy. Dig Dis Sci. 2022 Sep;67(9):4549-4556. doi: 10.1007/s10620-021-07316-4. Epub 2021 Dec 2. PMID 34859313
- [Background] Di Mitri R, Mocciaro F, Antonini F, Scimeca D, Conte E, Bonaccorso A, Scibetta N, Unti E, Fornelli A, Giorgini S, Binda C, Macarri G, Larghi A, Fabbri C. Stylet slow-pull vs. standard suction technique for endoscopic ultrasound-guided fine needle biopsy in pancreatic solid lesions using 20 Gauge Procore needle: A multicenter randomized trial. Dig Liver Dis. 2020 Feb;52(2):178-184. doi: 10.1016/j.dld.2019.08.023. Epub 2019 Oct 7. PMID 31601535
- [Background] Fujita A, Ryozawa S, Tanisaka Y, Ogawa T, Saito Y, Katsuda H, Miyaguchi K, Yasuda M, Araki R, Mashimo Y, Tashima T, Nakano Y, Terada R, Jinushi R, Mizuide M. Comparison of Fork-tip and Franseen needles for endoscopic ultrasound-guided fine-needle biopsy in pancreatic solid lesions: A propensity-matched analysis. DEN Open. 2022 Jun 28;3(1):e147. doi: 10.1002/deo2.147. eCollection 2023 Apr. PMID 35898843